CLINICAL TRIAL: NCT06243315
Title: A Prospective, Multicenter, Post-marketing Clinical Follow-up Research to Evaluate the Long-term Safety of Ellansé-S Dermal Filler Made of PCL Microspheres for the Correction of Moderate-to-severe Nasolabial Folds
Status: Enrolling by invitation | Type: Observational
Sponsor: AQTIS Medical B.V. (Other)
Responsible Party: Sponsor
Other Study IDs: Ellansé-S
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Moderate-to-severe Nasolabial Folds (3-4 Level of WSRS Scores) on Both Sides of the Face

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Ellansé-S — It is indicated for subcutaneous implantation to correct moderate-to-severe NLFs

SUMMARY:
This research is intended to evaluate the long-term safety of Ellansé-S PCL dermal filler for the correction of moderate-to-severe NLFs.

374 subjects. This clinical trial is designed as a prospective, multicenter, post-marketing clinical follow-up trial to evaluate the long-term safety of the investigational product, dermal filler made of PCL microspheres, for the correction of moderate-to-severe NLFs

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and above;
2. Subjects with moderate-to-severe nasolabial folds (3-4 level of WSRS scores) on both sides of the face
3. Intended to be treated with PCL microsphere filler;
4. Voluntarily participate in this test, cooperate with follow-up, and sign an informed consent form

Exclusion Criteria:

1. Obvious acne scar, pigmentation, active infection, inflammation, tumor, precancerous lesion or unhealed wound in the intended injection area;
2. Patients who have used permanent fillers (PMMA, hydrogel polymer, liquid silicone for injection, polyvinyl alcohol (PVA), bone cement, autologous fat, etc.) for nasolabial groove injection;
3. Patients who have received semi-permanent fillers (polycaprolactone, L-polylactic acid, hydroxyapatite, platelet-rich plasma, etc.) injection treatment in nasolabial sulch area in the past 24 months;
4. Patients who have received temporary fillers (hyaluronic acid, collagen, etc.) injection treatment in nasolabial groove in the past 12 months;
5. Patients who have received botox injection treatment in nasolabial sulci in the past 6 months;
6. The nasolabial groove has been treated with beauty plastic, focused ultrasound, chemical stripping, photoelectric (laser, photon, radio frequency) in the past 3 months;
7. Use of hormones or immunosuppressants within the past 1 month;
8. Subjects who have used anticoagulants in the last 2 weeks;
9. Subjects with a history of crabfoot, hyperplastic scars or cicatricial constitution;
10. Subjects with active sepsis;
11. Subjects with coagulation dysfunction;
12. Subjects with autoimmune diseases;
13. Allergic to polycaprolactone or known product ingredients;
14. Pregnant, pregnant and lactating subjects;
15. Participated in other clinical trials in the past 30 days;
16. Other situations determined by the researcher to be unsuitable for participation in this study;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This research will prospectively enroll and follow up all eligible subjects aged 18 years and older with moderate-to-severe NLFs.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
MAEs | 1 month,6 months,1 year, 2 years,3years,4years,5years
  The incidence of MAEs associated with the investigational product will be collected for all visits

SECONDARY OUTCOMES:
AE/SAE | 1 month,6 months,1 year, 2 years,3years,4years,5years
  The incidence of AE/SAE will be collected for all visits.
Improvement of WSRS scores | 1 month,6 months,1 year, 2 years
  During screening visits and postoperative follow-up, investigators will use digital cameras to take standardized digital photos of the subjects on both sides. Based on the severity of the nasolabial folds on both sides of the subjects, the improvement of WSRS scores of the nasolabial folds at 1 month 1, 6 months, 1 year, and 2 years postoperative will be calculated compared to the baseline. Please refer to the appendix for the scoring criteria.
GAIS scores after injection treatment | 1 month,6 months,1 year, 2 years
  Scores on the General Aesthetic Improvement Scale (GAIS) will be collected on both sides of the face at postoperative visit points (1 month postoperative , 6 months postoperative, 1 year postoperative, and 2 years postoperative) based on images obtained from standardized postoperative photographs. Please refer to the appendix for the scoring criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Second People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No